CLINICAL TRIAL: NCT05978453
Title: Blood Pressure Monitor#Model#BP7# Clincial Test
Brief Title: Blood Pressure Monitor Clinical Test (Cuff Range: 13.5cm-22cm)
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: Andon Health 11
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2022-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Subject use both BP7 Wrist Automatic Electronic BPM and mercury sphygmomanometers

SUMMARY:
The purpose of this study is to verify the accurancy of the blood pressure monitor device.

Cuff size of arm circumference: 13.5cm- 22cm.

ELIGIBILITY:
Inclusion Criteria:

* Normal blood pressure and hypertensive patients over 12 years old

Exclusion Criteria:

* Patients with serious arrhythmias or a high frequency of arrhythmias
* pregnant woman
* Other investigators believe that it is not suitable to participate in this clinical trial

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Normal blood pressure and hypertensive patients over 12 years old
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
blood pressure monitor accurancy | 30 minutes
  All the test results of the electronic blood pressure monitor is within the accuracy creteria, with the merury sphygmomanometer as control

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No